CLINICAL TRIAL: NCT06179472
Title: Infant Survival and Long-term Outcome Following Fetoscopic Endoluminal Tracheal Occlusion in Severe Left and Right Congenital Diaphragmatic Hernia, A Phase III Trial
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Mercy Hospital Kansas City (Other)
Collaborators: University of Wisconsin, Madison (Other); NAFTNet FETO Consortium (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00003414
Record Dates: First submitted 2023-11-27; First posted 2023-12-22 (Actual); Last update posted 2025-11-14 (Actual); Status verified 2025-11

CONDITIONS: Congenital Diaphragmatic Hernia
MeSH Terms: conditions — Hernias, Diaphragmatic, Congenital

STUDY DESIGN:
Intervention Model Description: Comparison of outcomes between patients who elect to receive the intervention versus those that do not in the specified time-frame
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Balloon Arm (Experimental): Participants who consent to the insertion and the removal of the Balt GOLDBAL2 Balloon.
  Interventions: Device: BALT GOLDBAL2 Balloon
- No Treatment (No Intervention): Patients who have been diagnosed with severe CDH at our site but choose not to participate in the study.

INTERVENTIONS:
Device: BALT GOLDBAL2 Balloon — Placement and retrieval of the GOLDBALLOON Detachable Balloon for severe CDH
  Arms: Balloon Arm

SUMMARY:
The purpose of the study is to determine the infant survival and long-term effects of performing Fetoscopic Endoluminal Tracheal Occlusion (FETO) surgery and removal of the BALT Goldbal2 balloon at Children's Mercy Hospital. We hypothesize that FETO balloon placement may increase survival and decrease morbidity when compared to standard prenatal care for the treatment of severe left or right congenital diaphragmatic hernia (CDH).

DETAILED DESCRIPTION:
FETO is an un-blinded non-randomized two arm feasibility and efficacy study being conducted at Children's Mercy Hospital.

Potential subjects will be identified from the patient's standard of care prenatal evaluation for CDH at Children's Mercy Hospital, which includes the following:

* Comprehensive obstetrical ultrasound examination including documentation of cervical length, gestational age, biometry, liver herniation, hepatic vasculature, sonographic lung volume, amniotic fluid level, membrane status, and lung-to-head circumference ratio (LHR) calculation.
* Fetal echocardiography to evaluate for structural cardiac anomalies
* Fetal Magnetic resonance imaging (MRI) 24 - 26 weeks gestation to confirm fetal liver herniation, calculate total fetal lung volume (TFLV) and Observed/Expected total fetal lung volume (O/E TFLV).
* Maternal history including demographics, physical examination, vital signs, height and weight
* Laboratory tests, including microarray and karyotype via amniocentesis
* Review of concomitant medications
* Psychosocial evaluation with a social worker and/or health psychologist.

Eligibility Review and Informed Consent Process

The Principal Investigator and member of the study team will review the informed consent document with eligible patients. This includes the following:

* Description of study rationale and design as well as explicit description of the experimental nature of the intervention
* Description and explanation in detail of the procedures
* Review of Inclusion/Exclusion criteria
* Psychosocial evaluation to identify family support and possible confounding social issues
* Patient Education including: CDH description, prenatal and neonatal development, general expected outcomes and management options
* Review all objective risks, benefits and alternatives of FETO intervention
* Review of questions and assessment of patient's understanding of study procedures and requirements.

Research Procedures

* Clearance for surgery by anesthesia and the obstetrical staff
* Testing for human immunodeficiency virus (HIV), Hepatitis B, Hepatitis C, if unable to obtain from referring physician
* A three-person panel of maternal-fetal subject matter experts, along with the Primary Investigator, will act as an Enrollment Oversight Committee and review all inclusion/exclusion source documentation and provide approval for subject enrollment prior to commencement of the FETO procedure.

Intervention Phase

The study procedure phase includes FETO surgery (balloon placement), weekly or biweekly monitoring after surgery, and balloon removal.

FETO Surgery - Research

* Physical examination including weight, laboratory tests, review of medications
* FETO will be completed at 27 weeks 0 days - 29 weeks 6 days gestation for those with an O/E LHR of <30%; for left-sided, and completed at 27 weeks 0 days to 29 weeks 6 days gestation for those with an O/E LHR of <45% in right-sided CDH.
* The procedure will be completed under ultrasound guidance and prophylactic tocolysis using nifedipine and vaginal progesterone suppository for the duration of pregnancy as well as potential addition of other tocolytics on an as-needed bases per standard maternal-fetal medicine protocols. Fetal analgesia and immobilization will consist of fentanyl, atropine and rocuronium.
* A 10 Fr trocar, 1.3mm fetoscope within a 3.0mm sheath (Karl Storz, Tuttlingen, Germany), and a detachable balloon occlusion (BALTACCI-BDPE, Balt, Montmorency, France) system will be used.
* Tocolysis with nifedipine, 20 mg every 6 hours for tocolysis as well as 100 mg vaginal progesterone suppository nightly for the duration of pregnancy, per the FDTC postoperative workflow for other fetoscopic procedures. Breakthrough contractions treated with Indomethacin and IV Magnesium sulfate, per maternal-fetal medicine guidelines. Subjects may be discharged following successful tocolysis for breakthrough contractions on oral nifedipine, 10-20 mg orally every 6 hours in addition to vaginal progesterone suppository for the duration of pregnancy.
* Serial measurements of sonographic lung volume and O/E LHR and evaluation for balloon location will begin 24-48 hours following surgery and continue throughout pregnancy by ultrasound evaluation until balloon removal.
* The expected hospital course is 24-48 hours; however it is possible that the subject will be hospitalized for complications or preterm labor. The subject will then be discharged to a nearby accommodation at the Ronald McDonald House of Kansas City, Missouri.
* The subject and support person will be required to reside within 30 minutes of Children's Mercy Hospital in anticipation of balloon removal.
* Subjects will be on modified bed rest for the first 2 weeks post discharge but subsequently allowed to graduate to moderate activity if the uterus is quiescent.
* Assess for possible adverse events/serious adverse events.

Weekly Check-ups (Balloon Insertion to Removal/delivery)

Standard of Care Procedures:

* Laboratory tests (if clinically indicated)
* Biophysical profiles will be performed weekly beginning at 32 weeks gestation
* Physical exam, including weight, review of medications
* Fetal ultrasounds weekly after balloon insertion until delivery

  * Ultrasounds performed weekly after balloon placement will consist of scans done for purposes of monitoring post-procedure status of the pregnancy. This includes observation of fetal heart rate, amniotic fluid levels, rule-out chorioamniotic membrane separation, signs of rupture of membranes, proper balloon placement, response to balloon placement, such as O/E LHR, and fetal surveillance, such as Biophysical Profile.

Research Procedures:

• Assessment of possible adverse events/serious adverse events

Pre-Op Balloon Removal between 32 weeks 0 days and 34 weeks 6 days- Research

* Medical record history and review
* Physical examination including weight, laboratory tests, review of medications
* Vitals signs, including blood pressure, temperature, weight
* Ultrasound - measurements of sonographic lung volume & O/E LHR, measurements of amniotic fluid level and membrane status
* Fetal MRI will be performed to evaluate TFLV and O/E TFLV the week of planned balloon removal (typically 5 weeks after placement)
* Fetal echocardiogram
* Clearance for surgery by anesthesia and the obstetrical staff. Anesthesia regional (spinal or epidural) in preparation for possible emergent delivery.
* Maternal corticosteroids will be administered 48 hours prior to removal of balloon occlusion
* Tocolysis administered - nifedipine 20 mg preoperatively and then every 6 hours for 48 hours. Breakthrough contractions treated with increased dose of nifedipine, Indomethacin or IV Magnesium sulfate, as per maternal-fetal medicine protocols.
* Assess for possible adverse events/serious adverse events

Removal of Balloon - Research

Fetoscopic removal of the balloon occlusion will be performed at 34 weeks 0 days to 34 weeks 6 days gestation.

The maximum duration of balloon implantation, if placed at 27 weeks 0 days and removed in the 34th week, is 7 weeks. For those balloons placed later in gestation or removed earlier electively or emergently the duration will be shorter.

* Pre-operative ultrasound, morning of procedure (standard of care, (SOC))
* Procedure - attempted US guided percutaneous needle puncture through maternal abdomen using 20-gauge needle
* Procedure - if needle aspiration unsuccessful, fetoscopic removal of balloon
* Assessment for possible adverse events/serious adverse events.

Delivery

Planned delivery will occur around 39 weeks.

Standard of Care Procedures:

* Surfactant will be administered if balloon is removed at the time of delivery, at delivery less than 34 weeks, or if the baby is born less than 96 hours after FETO release.
* Delivery
* Standard postnatal care
* For preterm labor before the balloon has been removed, the pregnant person will be admitted for tocolysis, maternal corticosteroids and attempt to maintain pregnancy.
* Laboratory tests
* Review of medications
* For preterm labor before the balloon has been removed that cannot be controlled by tocolysis, delivery by Ex Utero Intrapartum Therapy (EXIT), if maternally safe, may be performed. Emergent EXIT algorithms used as standard practice for fetuses with obstructed airway from other causes initiated. Systems are already in place for mothers presenting in labor prior to planned EXIT delivery.
* For precipitous preterm labor or maternal indications when EXIT cannot be performed, and prior to balloon removal, delivery by Cesarean section may be performed followed by immediate bronchoscopy and establishment of airway.

Research Procedures:

• Assessment for possible adverse events/serious adverse events.

Ensuring Proper Balloon Removal

* When an endoscope is in contact with an inflated balloon, one may actually look through the balloon, hence be under the (false) impression that one looks in a patent airway. There are indications that it is not the case, such as flattening of the mucosa and stretching of the trachea. Also when withdrawing the endoscope, the contour and tail of the balloon become immediately obvious.
* Working with real time video-endoscopy seems recommendable. It allows more comfortable visualization and the entire team can monitor the procedure and interact with the operator. It allows also documentation (filming) for inclusion in the medical record.
* There are several purpose-designed instruments available, yet also the insertion fetoscope can be used for balloon retrieval. It may be wise to use the instruments one is most familiar with. However, all these purpose designed instruments we described, allow water irrigation, so that one can clear debris and judge about the status of the airways
* There is also a high-fidelity training model that can be used for training and re-training.
* When one removes the balloon on placental circulation and there is no fetal distress, one has all the time to control the entire process of establishing airways. It is recommended to take the time to remove the balloon (or if punctured all fragments), suction and clear the airways, intubate and start ventilation while still on the cord. Only when positive signs of open and functional airways (including excursion of the chest and oxygenation signs) the cord should be clamped.

Follow-up Phase

The follow-up phase will be conducted from birth to 36 months of age. A resuscitation team from neonatology and pediatric surgery will be present at the delivery. A standard protocol will be utilized for postnatal care.

The results of Standard of Care Procedures, if performed, will be used for the research study and will be collected at time of birth, 6 months, 12 months, 24 months and 36 months (± 1 month). Extracted data from the electronic medical record (EMR) may include the following:

* Use of ECMO (type, timing, duration, ability to wean)
* Normalization of pulmonary vascular resistance. Utilization of pulmonary vasodilators (e.g., inhaled nitric oxide, sildenafil) per NICU and pediatric intensive care unit (PICU) guidelines.
* Bronchoscopy prior to initial discharge to document presence or absence of tracheomalacia (performed on a symptomatic basis only).
* Brain imaging - Head MRI
* Audiology examination
* Pulmonary function testing (PFT)
* Chest radiograph
* Physical exam and interim medical history
* Echocardiographic assessments

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated informed consent form
* Stated willingness to comply with all study procedures and availability (meets psychosocial criteria below) for the duration of the study
* Pregnant persons age 18 years and older
* Singleton pregnancy
* Absence of life-limiting genetic anomalies on microarray or karyotype on amniocentesis. Results by fluorescence in situ hybridization (FISH) will be acceptable if the patient is > 26 weeks gestation
* Fetal echocardiogram with changes expected with CDH and no major structural cardiac defects (small ventricular septal defect (VSD)/atrial septal defect (ASD) may be included as they will not alter outcome and are not life-limiting)
* Left or Right CDH with liver up without presence of concomitant life-limiting anomalies.
* Gestational age for Left-CDH at enrollment prior to 29 weeks plus 6 days for O/E LHR <30%; for Right-CDH with O/E LHR <45% gestational age at enrollment prior to 29 weeks plus 6 days.
* Meets psychosocial criteria
* Willing to reside within 30 minutes of Children's Mercy Hospital Fetal Health Center and ability to maintain follow up appointments
* Patient has a support person (e.g. spouse, partner, friend, or parent) that is available to stay with her for the duration of the pregnancy.
* Willing to comply with restrictions of daily living including inability to exercise, have intercourse or return to work.

Exclusion Criteria:

* Pregnant persons < 18 years of age
* Multi-fetal pregnancy
* Rubber latex allergy
* History of preterm labor, cervix shortened (<15mm at enrollment or within 24 hours of FETO balloon insertion procedure) or uterine anomaly strongly predisposing to preterm labor, placenta previa
* Psychosocial ineligibility precluding consent:

  * Inability to reside within 30 minutes of Children's Mercy Hospital Fetal Health Center until balloon removal or delivery (if clinically indicated)
  * Patient does not have a support person (e.g., spouse, partner, parent) available to stay with the patient until balloon removal or duration of the pregnancy (if clinically indicated)
  * Adult unable to consent
  * Prisoners
  * Social work or health psychology will meet with each patient to evaluate the social situation and support system. Identifiable issues of social instability or compliance with the protocol will exclude the patient as a potential candidate.
* Bilateral CDH, isolated left-sided with O/E LHR ≥30% (measured at 18 weeks 0 days to 29 weeks 5 days) as determined by ultrasound, isolated right-sided CDH with O/E LHR ≥45% (measured at 18 years 0 days to 29 weeks 5 days) as determined by ultrasound.
* Additional life-limiting fetal anomaly by ultrasound, MRI or echocardiogram that may affect outcome. These include chromosomal or anatomic abnormalities, associated anomalies recognized to alter survival prognosis (i.e., CDH and severe congenital heart disease) or presence of an underlying genetic syndrome (e.g., Fryns). No cases will be removed post hoc if abnormalities are discovered in the course of post-operative monitoring.
* Patient contraindication to fetoscopic surgery or severe medical condition in pregnancy
* History of incompetent cervix with or without cerclage
* Placental abnormalities (previa, abruption, accreta) known at the time of enrollment
* Pregnant person-fetal Rh isoimmunization, Kell sensitization or neonatal alloimmune thrombocytopenia affecting the current pregnancy
* Pregnant person tests positive for HIV, Hepatitis-B, Hepatitis-C. Due to of the increased risk of transmission to the fetus during maternal-fetal surgery the patient must test negative for these conditions prior to enrollment.
* Uterine anomaly such as large or multiple fibroids or mullerian duct abnormality
* There is no safe or technically feasible fetoscopic approach to balloon placement
* Participation in another intervention study that influences maternal and fetal morbidity and mortality or participation in this trial in a previous pregnancy.
* Patient refusal to receive blood products
* Additional major anomaly or abnormality that would prevent successful FETO, per discretion of the Principal Investigator

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-04-14 (Actual); Primary Completion 2031-01-01 (Estimated); Study Completion 2032-01-01 (Estimated)

PRIMARY OUTCOMES:
Infant survival | Birth to 24 months
  Infant survival will be measured from delivery to discharge, at 6, 12, and 24 months of age.
Number of occurrences and severity of pulmonary hypertension | Birth to 6 months
  Recording the occurrence of severe pulmonary hypertension based on echocardiogram
Use of Extracorporeal Membrane Oxygenation (ECMO) support | Birth to 6 months
  Number of infants requiring ECMO support

SECONDARY OUTCOMES:
Change in fetal lung growth | The first ultrasound within 1 week after balloon removal (balloon removal ideally at 34 weeks gestation)
  Prenatal ultrasound will measure the observed-to-expected lung to head ratio (o/e LHR) at weekly visits while the balloon is in place and after balloon removal. Fetal lung growth will be calculated as the difference between the o/e LHR pre-balloon placement and the o/e LHR after balloon removal.
Maternal Complications | Up to 4-6 weeks post-partum
  Complications during pregnancy, delivery, and first post-partum visit to include: preterm labor, premature rupture of membranes (PROM), preterm premature rupture of membranes (PPROM), oligohydramnios, polyhydramnios, placental abruption, chorioamnionitis, and other infection.
Gestational age at delivery | At the time of delivery
  Gestational age at delivery will be recorded.
Number of infants requiring supplemental oxygen | Birth to 24 months
  Supplemental oxygen requirement at time of discharge will be collected from medical chart review.
Number of days in neonatal intensive care unit (NICU) / pediatric intensive care unit (PICU) | Birth to 1 year
  Number of days that the neonate requires admission to the NICU/PICU

CONTACTS AND LOCATIONS:
Overall Officials: Inna Lobeck, Principal Investigator — Physician
Locations (1):
- Children's Mercy Hospital, Kansas City, Missouri, United States

IPD SHARING:
Plan to Share IPD: No